CLINICAL TRIAL: NCT02156466
Title: Multicenter, Phase I, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety, Tolerability, Immunogenicity, Pharmacokinetics, Pharmacodynamics and Efficacy of Multiple Ascending Doses of Subcutaneous MSB0010841 (Anti-IL17A/F Nanobody) in Male and Female Subjects With Moderate to Severe Psoriasis
Brief Title: Multiple Ascending Dose Trial of MSB0010841 (Anti-IL17A/F Nanobody) in Psoriasis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200574-003; 2013-005436-18 (EudraCT Number)
Record Dates: First submitted 2014-05-23; First posted 2014-06-05 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; MSB0010841; Anti-IL17A/F Nanobody; M1095
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- MSB0010841 30 mg (Experimental)
  Interventions: Drug: MSB0010841
- MSB0010841 60 mg (Experimental)
  Interventions: Drug: MSB0010841
- MSB0010841 120 mg (Experimental)
  Interventions: Drug: MSB0010841
- MSB0010841 240 mg (Experimental)
  Interventions: Drug: MSB0010841
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MSB0010841 — MSB0010841(Anti- IL-17A/F Nanobody) will be administered at a dose of 30 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
  Other Names: Anti-IL-17A/F Nanobody; M1095
  Arms: MSB0010841 30 mg
Drug: MSB0010841 — MSB0010841 will be administered at a dose of 60 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
  Other Names: Anti-IL-17A/F Nanobody; M1095
  Arms: MSB0010841 60 mg
Drug: MSB0010841 — MSB0010841 will be administered at a dose of 120 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
  Other Names: Anti-IL-17A/F Nanobody; M1095
  Arms: MSB0010841 120 mg
Drug: MSB0010841 — MSB0010841 will be administered at a dose of 240 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
  Other Names: Anti-IL-17A/F Nanobody; M1095
  Arms: MSB0010841 240 mg
Drug: Placebo — Placebo matched to MSB0010841 will be administered as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
  Arms: Placebo

SUMMARY:
This is a multicenter, Phase 1, randomized, double-blind, placebo-controlled trial in subjects with moderate to severe psoriasis to assess the safety, tolerability, immunogenicity, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of multiple subcutaneous ascending doses of MSB0010841 (Anti-interleukin-17A/F [Anti-IL-17A/F] Nanobody).

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis for at least 6 months before screening
* Greater than or equal to (>=) 10% of BSA with plaques
* Psoriasis Area and Severity Index (PASI) >=12
* Static Physician's Global Assessment (sPGA) >=3 (where scores range from 0 [clear of disease] to 5 [severe disease]) at the screening and baseline visits
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Any condition, including protocol-specified laboratory findings and findings in the medical history or in the pre-trial assessments which in the Investigator's opinion constitutes a risk or a contraindication for the subject's participation in the trial or that could interfere with the trial objectives, conduct or evaluation
* Currently having a form of non-plaque psoriasis as specified in the protocol
* Drug induced psoriasis
* Biological treatments as specified in the protocol, within 3 months prior to Day 1
* Systemic immunosuppressants or phototherapy as specified in the protocol, within 1 month prior to Day 1
* Use of anti-coagulant medications and/or antiplatelet medications as defined in the protocol
* Use of aspirin as defined in the protocol
* Topical corticosteroid treatments other than low-strength or lower-mid strength corticosteroids on the face, scalp, axillae, and/or groin within 1 month prior to Day 1
* Any previous treatment with an agent targeting interleukin (IL)-17, IL-12 and/or IL-23 as specified in the protocol
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 41 subjects were randomized in the trial and included in the Safety analysis set.
Groups:
- MSB0010841 30 mg: MSB0010841 (Anti-Interleukin [IL]-17A/F Nanobody) was administered at a dose of 30 milligram (mg) as subcutaneous (SC) injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
- MSB0010841 60 mg: MSB0010841 was administered at a dose of 60 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
- MSB0010841 120 mg: MSB0010841 was administered at a dose of 120 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
- MSB0010841 240 mg: MSB0010841 was administered at a dose of 240 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
- Placebo: Placebo matched to MSB0010841 was administered as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
Period: Overall Study
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Started | 8 | 8 | 8 | 9 | 8
Completed | 8 | 8 | 7 | 7 | 8
Not Completed | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Quantiferon Positivity | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all 41 subjects who received at least 1 dose of investigational medicinal product (IMP) (MSB0010841 or placebo).
Groups:
- MSB0010841 30 mg: MSB0010841 (Anti- IL-17A/F Nanobody) was administered at a dose of 30 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
- Total: Total of all reporting groups
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (13.24) | 42.1 (19.57) | 43.8 (13.59) | 44.8 (15.65) | 46.1 (14.57) | 45.1 (14.87)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 1 | 2 | 6
  Male | 7 | 8 | 6 | 8 | 6 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence which does not necessarily have a causal relationship with this the study drug. An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. TEAEs were the AEs occurring or worsening after treatment administration.
Time Frame: Baseline up to Day 85
Population: Safety analysis set included all 41 subjects who received at least 1 dose of IMP (MSB0010841 or placebo).
Measure: Number; unit: subjects
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
subjects | 6 | 5 | 5 | 6 | 6

2. Primary Outcome: Number of Subjects With Local Injection Site Reactions (ISRs)
Description: The injection site was assessed by the Principal Investigator (PI) or his/her designee for local reactions such as redness, swelling, indurations or bruising, and by the subject for itching. Redness and bruising were scaled as None (no visible redness or bruising present); Mild (less than or equal to [<=] 2.0 centimeters [cm] redness or bruising area); Moderate (greater than [>] 2 to <=5.0 cm redness or bruising area); Severe (>5.0 cm redness or bruising area). Swelling was scaled as None (no swelling detected); Mild (palpable 'firmness' only); Moderate (<= 4 cm swelling); Severe (>4 cm swelling). Induration was scaled as None (no induration); Mild (able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up); Moderate (able to slide skin, unable to pinch skin); Severe (unable to slide or pinch skin). Itching was scaled as No itching; Mild itching; Moderate itching and Severe itching. Subjects who reported any of the local ISRs were reported.
Time Frame: Day 1, 2,8, 15, 16, 22, 29, 30, 36, 43
Population: Safety analysis set included all 41 subjects who received at least one dose of IMP (MSB0010841 or placebo). Here "n" signifies those subjects who were evaluable for the specified injection site reaction. Subjects may be represented in more than 1 category.
Measure: Number; unit: subjects
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
subjects
  Day 1 Bruising: none (n=8,8,8,9,8) | 8 | 8 | 8 | 9 | 8
  Day 1 Indurations: none (n=8,8,8,9,8) | 8 | 8 | 7 | 9 | 8
  Day 1 Indurations: mild (n=8,8,8,9,8) | 0 | 0 | 1 | 0 | 0
  Day 1 Itching: none (n=8,8,8,9,8) | 8 | 8 | 8 | 8 | 9
  Day 1 Itching: mild (n=8,8,8,9,8) | 0 | 0 | 0 | 1 | 0
  Day 1 Redness: none (n=8,8,8,9,8) | 8 | 7 | 8 | 8 | 6
  Day 1 Redness: mild (n=8,8,8,9,8) | 0 | 1 | 0 | 1 | 2
  Day 1 Swelling: none (n=8,8,8,9,8) | 8 | 7 | 8 | 9 | 8
  Day 1 Swelling: mild (n=8,8,8,9,8) | 0 | 1 | 0 | 0 | 0
  Day 2 Bruising: none (n=8,8,8,9,8) | 5 | 8 | 8 | 9 | 8
  Day 2 Bruising: mild (n=8,8,8,9,8) | 3 | 0 | 0 | 0 | 0
  Day 2 Indurations: none (n=8,8,8,9,8) | 8 | 8 | 8 | 9 | 8
  Day 2 Itching: none (n=8,8,8,9,8) | 8 | 8 | 8 | 9 | 8
  Day 2 Redness: none (n=8,8,8,9,8) | 8 | 8 | 8 | 9 | 8
  Day 2 Swelling: none (n=8,8,8,9,8) | 8 | 8 | 8 | 9 | 8
  Day 8 Bruising: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 8 Indurations: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 8 Itching: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 8 Redness: none (n=8,8,8,8,8) | 7 | 8 | 8 | 8 | 8
  Day 8 Redness: mild (n=8,8,8,8,8) | 1 | 0 | 0 | 0 | 0
  Day 8 Swelling: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 15 Bruising: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 15 Indurations: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 15 Itching: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 15 Redness: none (n=8,8,8,8,8) | 8 | 7 | 7 | 8 | 8
  Day 15 Redness: mild (n=8,8,8,8,8) | 0 | 1 | 0 | 0 | 0
  Day 15 Redness: moderate (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 15 Swelling: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 16 Bruising: none (n=8,8,8,8,8) | 8 | 7 | 8 | 7 | 8
  Day 16 Bruising: mild (n=8,8,8,8,8) | 0 | 1 | 0 | 1 | 0
  Day 16 Indurations: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 16 Itching: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 16 Redness: none (n=8,8,8,8,8) | 7 | 8 | 8 | 8 | 8
  Day 16 Redness: mild (n=8,8,8,8,8) | 1 | 0 | 0 | 0 | 0
  Day 16 Swelling: none (n=8,8,8,8,8) | 8 | 8 | 7 | 8 | 8
  Day 16 Swelling: mild (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 22 Bruising: none (n=8,8,8,8,8) | 8 | 8 | 8 | 7 | 8
  Day 22 Bruising: mild (n=8,8,8,8,8) | 0 | 0 | 0 | 1 | 0
  Day 22 Indurations: none (n=8,8,8,8,8) | 8 | 8 | 7 | 8 | 8
  Day 22 Indurations: severe (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 22 Itching: none (n=8,8,8,8,8) | 7 | 8 | 8 | 8 | 8
  Day 22 Itching: mild (n=8,8,8,8,8) | 1 | 0 | 0 | 0 | 0
  Day 22 Redness: none (n=8,8,8,8,8) | 8 | 8 | 7 | 8 | 8
  Day 22 Redness: severe (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 22 Swelling: none (n=8,8,8,8,8) | 8 | 8 | 7 | 8 | 8
  Day 22 Swelling: severe (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 29 Bruising: none (n=8,8,8,7,8) | 8 | 8 | 8 | 7 | 8
  Day 29 Indurations: none (n=8,8,7,7,8) | 8 | 8 | 7 | 7 | 8
  Day 29 Itching: none (n=8,8,8,7,8) | 8 | 8 | 8 | 7 | 8
  Day 29 Redness: none (n=8,8,8,8,8) | 8 | 8 | 6 | 5 | 8
  Day 29 Redness: mild (n=8,8,8,8,8) | 0 | 0 | 2 | 2 | 0
  Day 29 Redness: moderate (n=8,8,8,8,8) | 0 | 0 | 0 | 1 | 0
  Day 29 Swelling: none (n=8,8,8,7,8) | 8 | 8 | 7 | 7 | 8
  Day 29 Swelling: mild (n=8,8,8,7,8) | 0 | 0 | 1 | 0 | 0
  Day 30 Bruising: none (n=8,8,8,7,8) | 8 | 8 | 7 | 6 | 8
  Day 30 Bruising: mild (n=8,8,8,7,8) | 0 | 0 | 1 | 1 | 0
  Day 30 Indurations: none (n=8,8,7,7,8) | 8 | 8 | 7 | 7 | 8
  Day 30 Itching: none (n=8,8,7,7,8) | 8 | 8 | 0 | 0 | 8
  Day 30 Redness: none (n==8,8,7,7,8) | 8 | 8 | 7 | 6 | 8
  Day 30 Redness: moderate (n=8,8,7,7,8) | 0 | 0 | 0 | 1 | 0
  Day 30 Swelling: none (n=8,8,7,7,8) | 8 | 8 | 7 | 7 | 8
  Day 36 Bruising: none (n=7,8,7,7,8) | 7 | 8 | 7 | 6 | 8
  Day 36 Bruising: mild (n=7,8,7,7,8) | 0 | 0 | 0 | 1 | 0
  Day 36 Indurations: none (n=8,8,7,7,7) | 8 | 8 | 7 | 7 | 7
  Day 36 Itching: none (n=7,8,7,6,8) | 7 | 8 | 7 | 6 | 8
  Day 43 Bruising: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 43 Indurations: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 43 Itching: none (8,8,8,8,8) | 8 | 8 | 8 | 8 | 8
  Day 43 Redness: none (n=8,8,8,8,8) | 8 | 8 | 7 | 8 | 8
  Day 43 Redness: moderate (n=8,8,8,8,8) | 0 | 0 | 1 | 0 | 0
  Day 43 Swelling: none (n=8,8,8,8,8) | 8 | 8 | 8 | 8 | 8

3. Primary Outcome: Amount of Pain at Injection Site Assessed By Visual Analog Scale (VAS)
Description: Subjects were asked to assess their severity of injection site pain on a 100 millimeter (mm) VAS, where 0 = no pain and 100 = worst possible pain. Mean of amount of pain was calculated for the subjects having a value > 0. Maximum values per subjects (over injection site areas) are used for counting the amount of pain at injection site. Maximum pain scores recorded among all participants analysed in each arm are reported for each time point.
Time Frame: Day 1, 2, 8, 15, 16, 22, 29, 30, 36, 43
Population: Safety analysis set included all 41 subjects who received at least one dose of IMP (MSB0010841 or placebo). Here "Number of subjects analyzed" signifies those subjects who were evaluable for this endpoint and "n" signifies those subjects who were evaluable at the specified time point.
Measure: Number; unit: mm
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 6 | 8 | 4 | 8
mm
  Day 1 (n=3,2,3,2,0) | 7 | 4 | 7 | 4 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 2 (n=1,1,1,1,0) | 1 | 1 | 1 | 1 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 8 (n=1,1,0,0,0) | 1 | 1 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 15 (n=2,1,3,0,0) | 5 | 3 | 7 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 16 (n=0,0,0,0,2) | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | 2
  Day 22 (1,0,1,0,0) | 11 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | 1 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 29 (n=1,1,1,0,0) | 3 | 2 | 2 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 30 (1,0,1,1,0) | 2 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | 1 | 1 | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 36 (n=0,0,0,0,0) | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point
  Day 43 (n=0,0,0,0,0) | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point | NA — Data could not be calculated as there were no subjects with amount of pain value of > 0 at the specified time point

4. Primary Outcome: Percentage of Subjects With Anti-MSB0010841 Binding Antibodies (Anti-Drug Antibodies [ADA])
Description: Data were presented for MSB0010841 combined group and placebo.
Time Frame: Baseline up to Day 85
Population: Safety analysis set included all 41 subjects who received at least one dose of IMP (MSB0010841 or placebo).
Measure: Number; unit: percentage of subjects
Groups:
- MSB0010841 Combined: All subjects who received MSB0010841 (Anti-IL-17A/F Nanobody) at a dose of 30 mg, 60 mg, 120 mg or 240 mg as subcutaneous (SC) injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks
Arm/Group | MSB0010841 Combined | Placebo
Number analyzed (Participants) | 33 | 8
percentage of subjects | 30.3 | 37.5

5. Primary Outcome: Levels of Anti-MSB0010841 Antibody Titers
Time Frame: Day 8, 15 (pre-dose), 22, 29 (pre-dose), 36, 43, 63 and 85
Population: All subjects who received placebo or MSB0010841 (30 mg, 60 mg, 90 mg or 240 mg) and had positive ADA titers before and/or after study drug administration were included in the analysis population.
Measure: Number; unit: log10titer
Groups:
- ADA Positive Subjects: All subjects who received placebo or MSB0010841 (30 mg, 60 mg, 90 mg or 240 mg) and had positive ADA titers before and/or after study drug administration.
Arm/Group | ADA Positive Subjects
Number analyzed (Participants) | 13
log10titer
  Day 8 Subject 1: Placebo | 3.68
  Day 8 Subject 2: Placebo | 3.68
  Day 8 Subject 3: Placebo | 3.68
  Day 8 Subject 4: MSB0010841 30 mg | 3.68
  Day 8 Subject 5: MSB0010841 30 mg | 0
  Day 8 Subject 6: MSB0010841 30 mg | 2.28
  Day 8 Subject 7: MSB0010841 60 mg | 0
  Day 8 Subject 8: MSB0010841 120 mg | 3.68
  Day 8 Subject 9: MSB0010841 120 mg | 4.38
  Day 8 Subject 10: MSB0010841 120 mg | 3.68
  Day 8 Subject 11: MSB0010841 120 mg | 4.38
  Day 8 Subject 12: MSB0010841 120 mg | 2.98
  Day 8 Subject 13: MSB0010841 240 mg | 2.98
  Day 15 (pre-dose) Subject 1: Placebo | 3.68
  Day 15 (pre-dose) Subject 2: Placebo | 3.68
  Day 15 (pre-dose) Subject 3: Placebo | 3.68
  Day 15 (pre-dose) Subject 4: MSB0010841 30 mg | 3.68
  Day 15 (pre-dose) Subject 5: MSB0010841 30 mg | 0
  Day 15 (pre-dose) Subject 6: MSB0010841 30 mg | 2.28
  Day 15 (pre-dose) Subject 7: MSB0010841 60 mg | 2.98
  Day 15 (pre-dose) Subject 8: MSB0010841 120 mg | 5.78
  Day 15 (pre-dose) Subject 9: MSB0010841 120 mg | 4.38
  Day 15 (pre-dose) Subject 10: MSB0010841 120 mg | 3.68
  Day 15 (pre-dose) Subject 11: MSB0010841 120 mg | 4.38
  Day 15 (pre-dose) Subject 12: MSB0010841 120 mg | 2.98
  Day 15 (pre-dose) Subject 13: MSB0010841 240 mg | 2.98
  Day 22 Subject 1: Placebo | 3.68
  Day 22 Subject 2: Placebo | 3.68
  Day 22 Subject 3: Placebo | 3.68
  Day 22 Subject 4: MSB0010841 30 mg | 3.68
  Day 22 Subject 5: MSB0010841 30 mg | 2.98
  Day 22 Subject 6: MSB0010841 30 mg | 2.98
  Day 22 Subject 7: MSB0010841 60 mg | 2.28
  Day 22 Subject 8: MSB0010841 120 mg | 2.98
  Day 22 Subject 9: MSB0010841 120 mg | 4.38
  Day 22 Subject 10: MSB0010841 120 mg | 3.68
  Day 22 Subject 11: MSB0010841 120 mg | 4.38
  Day 22 Subject 12: MSB0010841 120 mg | 2.98
  Day 22 Subject 13: MSB0010841 240 mg | 2.98
  Day 29 (pre-dose) Subject 1: Placebo | 3.68
  Day 29 (pre-dose) Subject 2: Placebo | 3.68
  Day 29 (pre-dose) Subject 3: Placebo | 3.68
  Day 29 (pre-dose) Subject 4: MSB0010841 30 mg | 2.98
  Day 29 (pre-dose) Subject 5: MSB0010841 30 mg | 0
  Day 29 (pre-dose) Subject 6: MSB0010841 30 mg | 2.98
  Day 29 (pre-dose) Subject 7: MSB0010841 60 mg | 2.28
  Day 29 (pre-dose) Subject 8: MSB0010841 120 mg | 3.68
  Day 29 (pre-dose) Subject 9: MSB0010841 120 mg | 3.68
  Day 29 (pre-dose) Subject 10: MSB0010841 120 mg | 3.68
  Day 29 (pre-dose) Subject 11: MSB0010841 120 mg | 4.38
  Day 29 (pre-dose) Subject 12: MSB0010841 120 mg | 2.98
  Day 29 (pre-dose) Subject 13: MSB0010841 240 mg | 2.98
  Day 36 Subject 1: Placebo | NA — Data were not assessed as no sample was collected at this time point
  Day 36 Subject 2: Placebo | 3.68
  Day 36 Subject 3: Placebo | 3.68
  Day 36 Subject 4: MSB0010841 30 mg | 2.98
  Day 36 Subject 5: MSB0010841 30 mg | 0
  Day 36 Subject 6: MSB0010841 30 mg | 2.98
  Day 36 Subject 7: MSB0010841 60 mg | 2.98
  Day 36 Subject 8: MSB0010841 120 mg | NA — Data were not assessed as no sample was collected at this time point
  Day 36 Subject 9: MSB0010841 120 mg | 3.68
  Day 36 Subject 10: MSB0010841 120 mg | 4.38
  Day 36 Subject 11: MSB0010841 120 mg | 4.38
  Day 36 Subject 12: MSB0010841 120 mg | 3.68
  Day 36 Subject 13: MSB0010841 240 mg | 2.98
  Day 43 Subject 1: Placebo | 2.98
  Day 43 Subject 2: Placebo | 3.68
  Day 43 Subject 3: Placebo | 3.68
  Day 43 Subject 4: MSB0010841 30 mg | 2.98
  Day 43 Subject 5: MSB0010841 30 mg | 0
  Day 43 Subject 6: MSB0010841 30 mg | 2.98
  Day 43 Subject 7: MSB0010841 60 mg | 2.28
  Day 43 Subject 8: MSB0010841 120 mg | 4.38
  Day 43 Subject 9: MSB0010841 120 mg | 3.68
  Day 43 Subject 10: MSB0010841 120 mg | 4.38
  Day 43 Subject 11: MSB0010841 120 mg | 3.68
  Day 43 Subject 12: MSB0010841 120 mg | 2.98
  Day 43 Subject 13: MSB0010841 240 mg | 2.98
  Day 63 Subject 1: Placebo | 3.68
  Day 63 Subject 2: Placebo | 3.68
  Day 63 Subject 3: Placebo | 3.68
  Day 63 Subject 4: MSB0010841 30 mg | 4.38
  Day 63 Subject 5: MSB0010841 30 mg | 0
  Day 63 Subject 6: MSB0010841 30 mg | 2.98
  Day 63 Subject 7: MSB0010841 60 mg | 2.28
  Day 63 Subject 8: MSB0010841 120 mg | 2.98
  Day 63 Subject 9: MSB0010841 120 mg | 3.68
  Day 63 Subject 10: MSB0010841 120 mg | 3.68
  Day 63 Subject 11: MSB0010841 120 mg | 3.68
  Day 63 Subject 12: MSB0010841 120 mg | 3.68
  Day 63 Subject 13: MSB0010841 240 mg | 2.98
  Day 85 Subject 1: Placebo | 3.68
  Day 85 Subject 2: Placebo | 3.68
  Day 85 Subject 3: Placebo | 3.68
  Day 85 Subject 4: MSB0010841 30 mg | 3.68
  Day 85 Subject 5: MSB0010841 30 mg | 0
  Day 85 Subject 6: MSB0010841 30 mg | 2.28
  Day 85 Subject 7: MSB0010841 60 mg | 2.28
  Day 85 Subject 8: MSB0010841 120 mg | 2.98
  Day 85 Subject 9: MSB0010841 120 mg | 3.68
  Day 85 Subject 10: MSB0010841 120 mg | 3.68
  Day 85 Subject 11: MSB0010841 120 mg | 2.98
  Day 85 Subject 12: MSB0010841 120 mg | 3.68
  Day 85 Subject 13: MSB0010841 240 mg | 2.98

6. Primary Outcome: Levels of Pre-existing Anti-MSB0010841 Antibody Titers
Time Frame: Pre-dose on Day 1
Population: as for outcome 5
Measure: Number; unit: log10titer
Arm/Group | ADA Positive Subjects
Number analyzed (Participants) | 13
log10titer
  Subject 1: Placebo | 2.98
  Subject 2: Placebo | 3.68
  Subject 3: Placebo | 3.68
  Subject 4: MSB0010841 30 mg | 2.98
  Subject 5: MSB0010841 30 mg | 0
  Subject 6: MSB0010841 30 mg | 0
  Subject 7: MSB0010841 60 mg | 0
  Subject 8: MSB0010841 120 mg | 2.98
  Subject 9: MSB0010841 120 mg | 5.08
  Subject 10: MSB0010841 120 mg | 3.68
  Subject 11: MSB0010841 120 mg | 3.68
  Subject 12: MSB0010841 120 mg | 2.98
  Subject 13: MSB0010841 240 mg | 0

7. Primary Outcome: MSB0010841 Serum Concentration Over Time After First Dose
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: PK analysis set included subjects who received first dose of MSB0010841 without protocol deviations affecting PK, and who provide evaluable PK data. Here "n" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 9
nanogram/milliliter (ng/mL)
  0 hour (n=8,8,8,9) | 12.6 (35.71) | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)
  6 hour (n=8,8,8,9) | 907.5 (523.16) | 2097.1 (1391.43) | 2315.5 (787.02) | 4858.8 (2326.35)
  12 hour (n=8,8,8,9) | 1793.3 (761.23) | 3339.6 (1671.29) | 4983.1 (1501.41) | 9780.3 (4698.97)
  24 hour (n=8,8,8,9) | 2788.4 (895.89) | 5047.8 (1600.25) | 9131.3 (2838.02) | 15357.6 (5295.18)
  32 hour (n=8,8,8,9) | 3037.3 (820.76) | 6028.1 (2269.66) | 11372.4 (3499.37) | 17135.2 (6032.66)
  72 hour (n=8,8,7,8) | 3190.4 (810.18) | 6492.9 (1472.29) | 11284.1 (2562.84) | 20536.6 (6716.38)
  96 hour (n=8,8,8,8) | 3155.8 (879.56) | 6423.8 (1824.46) | 11790.0 (3319.36) | 18732.9 (4670.66)
  168 hour (n=8,8,8,8) | 2665.5 (605.89) | 5179.5 (1126.74) | 10318.6 (2837.81) | 17761.9 (3072.48)
  336 hour (n=8,8,8,8) | 1704.3 (429.78) | 3951.0 (1353.92) | 6768.4 (2846.24) | 11605.8 (2065.58)

8. Primary Outcome: MSB0010841 Serum Concentration Over Time After Second Dose
Time Frame: 0 hours (pre-dose), 24, 72, 96, 168, 336 hours post-second dose (Day 15)
Population: PK analysis set included subjects who received active treatment (MSB0010841) without protocol deviations affecting PK, and who provide evaluable PK data. Here "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  0 hour | 1704.3 (429.78) | 3951.0 (1353.92) | 6768.4 (2846.24) | 11605.8 (2065.58)
  24 hour | 3808.0 (980.68) | 7268.9 (3771.98) | 15120.6 (3393.84) | 27664.8 (9231.41)
  72 hour | 4309.0 (1265.45) | 9095.5 (2115.16) | 17454.4 (4152.32) | 29902.4 (7523.13)
  96 hour | 4020.5 (923.65) | 8514.4 (1849.44) | 17081.4 (5056.17) | 29223.5 (8336.26)
  168 hour | 3517.8 (877.96) | 7180.4 (1705.24) | 14806.6 (5632.99) | 22972.5 (11219.87)
  336 hour | 2306.5 (588.50) | 4492.9 (1398.63) | 10468.9 (4376.75) | 16454.5 (4548.85)

9. Primary Outcome: MSB0010841 Serum Concentration Over Time After Third Dose
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
ng/mL
  0 hour | 2306.5 (588.50) | 4492.9 (1398.63) | 10417.7 (4724.84) | 16173.6 (4837.78)
  6 hour | 3483.9 (1566.88) | 6200.1 (1391.38) | 12725.0 (5573.11) | 20452.3 (6683.19)
  12 hour | 3557.9 (1004.43) | 8615.5 (3093.46) | 13361.0 (5959.26) | 26051.4 (8770.65)
  24 hour | 4533.3 (1178.14) | 9969.9 (2494.60) | 17523.1 (6140.31) | 33651.7 (11590.56)
  32 hour | 4934.5 (1256.47) | 10762.5 (2377.88) | 18634.9 (5713.14) | 38278.4 (13391.40)
  72 hour | 4936.0 (1387.50) | 10345.6 (4586.24) | 19813.1 (6381.27) | 37166.4 (10103.58)
  96 hour | 4994.9 (1448.53) | 9047.6 (2760.25) | 18260.1 (6602.90) | 33909.3 (10219.54)
  168 hour | 4368.1 (1201.56) | 7715.4 (3019.93) | 15585.3 (5625.65) | 31375.9 (6826.50)
  336 hour | 2680.5 (859.35) | 5602.1 (3057.34) | 12257.6 (7468.85) | 20011.9 (6248.98)
  504 hour | 1802.0 (505.42) | 3109.1 (1519.66) | 8610.6 (5991.68) | 12472.4 (4176.00)
  816 hour | 933.1 (376.76) | 1378.1 (834.66) | 4309.3 (4044.88) | 5064.6 (2070.93)
  1056 hour | 464.5 (257.13) | 658.5 (391.39) | 2599.7 (2937.08) | 2475.9 (1391.08)
  1344 hour | 244.8 (162.24) | 326.3 (230.87) | 1611.3 (2199.92) | 1345.7 (879.15)

10. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) Post First Dose of MSB0010841
Description: Area under the serum concentration-time curve (AUC) from time zero to the last sampling time point at which the concentration is at or above lower limit of quantification (LLOQ).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: PK analysis set included subjects who received active treatment (MSB0010841) without protocol deviations affecting PK, and who provide evaluable PK data. Here "Number of participants analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter (day*mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
day*microgram per milliliter (day*mcg/mL | 33.6 (28.0) | 69.3 (18.9) | 126.3 (28.5) | 216.5 (23.4)

11. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) Post Third Dose of MSB0010841
Description: Area under the serum concentration-time curve (AUC) from time zero to the last sampling time point at which the concentration is at or above LLOQ.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
day*mcg/mL | 93.7 (41.4) | 170.3 (39.5) | 371.7 (62.0) | 663.4 (31.1)

12. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUCtau) Post First Dose of MSB0010841
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (336 hours).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
day*mcg/mL | 32.4 (31.2) | 68.3 (16.4) | 114.6 (24.2) | 222.2 (19.6)

13. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero up to Time Tau (AUCtau) Post Third Dose of MSB0010841
Description: Area under the concentration-time curve from time zero up to time Tau, where Tau is the dosing interval (336 hours).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
day*mcg/mL | 54.2 (36.3) | 104.1 (33.9) | 203.2 (43.6) | 397.6 (27.1)

14. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC 0-inf) Post Third Dose of MSB0010841
Description: Area under the serum concentration-time curve from time zero to infinity (AUC0-inf). AUC0-infcalculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clast calc/λz, where Clast calc is the calculated concentration at the last sampling time point at which the measured concentration is at or above LLOQ and λz is the terminal rate constant determined from the terminal slope of the log transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
day*ug/mL | 97.6 (42.2) | 174.9 (39.9) | 392.6 (68.8) | 680.9 (32.2)

15. Primary Outcome: Observed Serum Concentration Immediately Before First Dose (Cpre) of MSB0010841
Description: The observed serum concentration immediately before the first dose.
Time Frame: Pre-dose (0 hours) on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
mcg/mL | 0.01 (0.036) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

16. Primary Outcome: Observed Serum Concentration Immediately Before Third Dose (Cpre) of MSB0010841
Description: The observed serum concentration immediately before the third dose.
Time Frame: Pre-dose (0 hours) on Day 29
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
mcg/mL | 2.31 (0.59) | 4.49 (1.40) | 10.42 (4.72) | 16.17 (4.84)

17. Primary Outcome: Minimum Concentration Observed (Cmin) During First Dosing Interval of MSB0010841
Description: The observed minimum serum concentration determined directly from the serum concentration-time profile of each subject.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
mcg/mL | 0.01 (0.036) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

18. Primary Outcome: Minimum Concentration Observed (Cmin) During Third Dosing Interval of MSB0010841
Description: The observed minimum serum concentration determined directly from the serum concentration-time profile of each subject.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
mcg/mL | 2.30 (0.60) | 4.34 (1.40) | 10.03 (4.95) | 16.17 (4.84)

19. Primary Outcome: Maximum Concentration Observed (Cmax) Post First Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
mcg/mL | 3.3 (28.4) | 7.4 (22.9) | 12.5 (25.6) | 20.8 (30.3)

20. Primary Outcome: Maximum Concentration Observed (Cmax) Post Third Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
mcg/mL | 5.14 (34.5) | 11.32 (29.7) | 19.74 (31.3) | 37.93 (32.2)

21. Primary Outcome: Average Concentration (Cav) Post First Dose of MSB0010841
Description: Cav was calculated by AUCtau/tau. Where tau is the dosing interval (336 hours).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
mcg/mL | 2.315 (31.2) | 4.881 (16.4) | 8.187 (24.2) | 15.868 (19.6)

22. Primary Outcome: Average Concentration (Cav) Post Third Dose of MSB0010841
Description: Cav was calculated by AUCtau/tau. Where tau is the dosing interval (336 hours).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
mcg/mL | 3.87 (36.3) | 7.44 (33.9) | 14.51 (43.6) | 28.40 (27.1)

23. Primary Outcome: Mean Residence Time (MRT0-t) Post First Dose of MSB0010841
Description: MRT is the average time at which the number of absorbed molecules reside in the body, after single-dose administration, and calculated as AUMC(0-t)/AUC(0-t) where AUMC(0-t) is area under the plasma concentration-time first moment curve from time zero to time t (336 hours) and AUC(0-t) is the area under the plasma concentration-time curve from time zero to tome t (336 hours).
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
day | 6.528 (3.6) | 6.691 (8.1) | 6.638 (5.7) | 6.771 (5.3)

24. Primary Outcome: Mean Residence Time (MRT0-t) Post Third Dose of MSB0010841
Description: as for outcome 23
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
day | 17.57 (11.2) | 15.68 (16.3) | 19.26 (32.0) | 16.38 (11.3)

25. Primary Outcome: Mean Residence Time of Drug in the Body From Time Zero Extrapolated to Infinity (MRT(0-inf) Post Third Dose of MSB0010841
Description: Mean residence time of drug in the body from time zero extrapolated to infinity, based on the last predicted concentration at tlast.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Groups:
- MSB0010841 30 mg: MSB0010841(Anti- IL-17A/F Nanobody) was administered at a dose of 30 mg as SC injection every other week (Day 1, Day 15 and Day 29) for a total duration of 6 weeks.
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
day | 17.57 (11.2) | 15.68 (16.3) | 19.26 (32.0) | 16.38 (11.3)

26. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) Post First Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour | 72.39 [23.9 to 97.4] | 71.68 [24.0 to 335.8] | 52.00 [32.0 to 96.2] | 72.23 [72.0 to 168.0]

27. Primary Outcome: Time to Maximum Observed Concentration (Tmax) Post Second Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 24, 72, 96, 168, 336 hours post-second dose (Day 15)
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour | 84.2 [72.0 to 97.5] | 72.0 [24.1 to 96.6] | 83.4 [71.8 to 168.0] | 72.0 [24.0 to 168.0]

28. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) Post Third Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
hour | 31.5 [6.0 to 95.8] | 31.0 [12.0 to 72.4] | 72.0 [31.8 to 72.5] | 72.0 [31.1 to 168.0]

29. Primary Outcome: Apparent Terminal Half-life (t1/2) Post Third Dose of MSB0010841
Description: Terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life is calculated by dividing the natural logarithm to the base e (Log e) multiplied by (*) 2/ λz, where 'λz' is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
day | 10.63 (17.3) | 10.50 (18.9) | 12.19 (27.9) | 10.25 (13.1)

30. Primary Outcome: Terminal Rate Constant (λz) Post Third Dose of MSB0010841
Description: Terminal rate constant was determined from the terminal slope of the logtransformed concentration curve using linear regression on terminal data points of the curve
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
1/hour | 0.00 (17.3) | 0.00 (18.9) | 0.00 (27.9) | 0.00 (13.1)

31. Primary Outcome: Apparent Clearance (CL/f) Post Third Dose of MSB0010841
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Apparent clearance after oral dose (CL/f) is influenced by the fraction absorbed.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
L/day | 0.55 (36.3) | 0.58 (33.9) | 0.59 (43.6) | 0.60 (27.1)

32. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) Post Third Dose of MSB0010841
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution during the terminal phase, calculated as Vz = Dose/AUC0-inf multiplied by elimination rate constant [λz]) following first dose and Dose/(AUCtau multiplied by λz) after third dose.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: PK analysis set included subjects who received active treatment (MSB0010841) without protocol deviations affecting PK, and who provide evaluable PK data. Here "Number of subjects analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
Liters | 8.49 (27.0) | 8.73 (38.6) | 10.39 (21.9) | 8.92 (18.8)

33. Primary Outcome: Percentage Peak-Trough Fluctuation (PTF) Post First Dose of MSB0010841
Description: The peak trough fluctuation within one dosing interval, calculated as PTF (%) = ([Cmax - Cmin]/Cav ) multiplied by 100
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1)
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
percentage fluctuation | 140.28 (3.9) | 152.47 (20.4) | 144.37 (13.0) | 135.89 (12.3)

34. Primary Outcome: Percentage Peak-Trough Fluctuation (PTF) Post Third Dose of MSB0010841
Description: The peak trough fluctuation within one dosing interval, calculated as PTF (%) = ([Cmax - Cmin]/Cav ) multiplied by 100
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 7 | 7
percentage fluctuation | 75.26 (8.5) | 95.65 (18.9) | 71.17 (33.1) | 76.03 (28.6)

35. Primary Outcome: Accumulation Ratio of Cmax (Racc (Cmax))
Description: Accumulation ratio for Cmax was calculated as Cmax, after third dose / Cmax, after first dose.
Time Frame: 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336 hours post-first dose (Day 1) and 0 hours (pre-dose), 6, 12, 24, 32, 72, 96, 168, 336, 504, 816, 1056, 1344 hours post-third dose (Day 29)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
ratio | 1.56 (17.9) | 1.52 (23.5) | 1.56 (34.1) | 1.81 (9.5)

36. Primary Outcome: Accumulation Ratio of AUC (Racc(AUC))
Description: Accumulation ratio for AUC, calculated as area under the serum concentration-time curve within one complete dosing interval at third dose divided by area under the serum concentration-time curve within one complete dosing interval at first dose.
Time Frame: as for outcome 35
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
ratio | 1.61 (15.9) | 1.50 (18.4) | 1.61 (27.4) | 1.83 (11.5)

37. Primary Outcome: Maximum Observed Concentration (Cmax) Post Second Dose of MSB0010841
Time Frame: 0 hours (pre-dose), 24, 72, 96, 168, 336 hours post-second dose (Day 15)
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
mcg/mL | 4.26 (32.7) | 9.06 (24.2) | 18.59 (23.1) | 30.98 (25.3)

38. Primary Outcome: Observed Serum Concentration Immediately Before Second Dose (Cpre) of MSB0010841
Description: The observed serum concentration immediately before second dose.
Time Frame: Pre-dose (0 hours) on Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
mcg/mL | 1.65 (30.2) | 3.74 (37.9) | 6.34 (38.3) | 11.44 (18.1)

39. Secondary Outcome: Percentage of Subjects With 50% or 75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: PASI: a physician assessed index that measured psoriasis severity and evaluated erythema, infiltration, and desquamation (scaling) on different body areas including the head, upper extremities, the trunk, and lower extremities. T Erythema, infiltration, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score. PASI score ranged from 0 to 72, with higher scores reflecting greater disease severity. PASI 50% or 75% was defined as the percentage of participants who achieved >=50 or 75% improvement in PASI score from Baseline.
Time Frame: Baseline up to Day 85
Population: Safety analysis set included all 41 subjects who received at least 1 dose of IMP (MSB0010841 or placebo).
Measure: Number; unit: percentage of subjects
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
percentage of subjects
  PASI-50 | 100 | 100 | 100 | 100 | 50
  PASI-75 | 88 | 100 | 100 | 100 | 0

40. Secondary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Day 43
Description: PASI: a physician assessed index that measured psoriasis severity and evaluated erythema, infiltration, and desquamation (scaling) on different body areas including the head, upper extremities, the trunk, and lower extremities. T Erythema, infiltration, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The total qualitative score (sum of erythema, thickness, and scaling scores) was multiplied by the degree of involvement for each anatomic region and then multiplied by a constant. These values for each anatomic region are summed to yield the PASI score. PASI score ranged from 0 to 72, with higher scores reflecting greater disease severity. PASI 50% or 75% was defined as the percentage of subjects who achieved >=50 or 75% improvement in PASI score from Baseline.
Time Frame: Baseline, Day 43
Population: Safety analysis set included all 41 subjects who received at least one dose of IMP (MSB0010841 or placebo).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
units on a scale
  Baseline | 16.91 (5.75) | 19.76 (4.79) | 23.35 (6.60) | 18.38 (6.07) | 25.49 (5.58)
  Change at Day 43 | -13.93 (4.76) | -17.99 (5.52) | -21.70 (8.52) | -16.68 (8.38) | -5.43 (7.04)

41. Secondary Outcome: Percentage of Subjects With Static Physician's Global Assessment (sPGA) Score of Minimal or Clear and With at Least 2 Level Reduction From Baseline
Description: The static Physician's Global Assessment (sPGA) scale rated the investigator's overall clinical assessment of a subjects plaque thickness, erythema, and scaling on a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (majority of plaques have severe thickness, erythema, and scale). To assign a sPGA score, the investigator examined all psoriatic lesions and assigned a severity score ranging from 0 to 5 for thickness, erythema, and scaling. Scores for thickness, erythema, and scaling are summed and the mean of these 3 scores equals the overall sPGA score. Overall sPGA score ranged from 0 to 5, where lower scores indicate clinical improvement. Percentage of subjects who achieved a sPGA rating of 0 (clear) or 1 (minimal) and had at Least 2 level reduction from Baseline score were reported.
Time Frame: Day 8, 15, 22, 29, 36, 43, 50, 85
Population: Safety analysis set included all 41 subjects who received at least one dose of IMP (MSB0010841 or placebo).
Measure: Number; unit: percentage of subjects
Groups:
- MSB0010841 30 mg: MSB0010841 was administered at a dose of 30 mg as SC injection every other week for a total duration of 6 weeks.
- MSB0010841 60 mg: MSB0010841 was administered at a dose of 60 mg as SC injection every other week for a total duration of 6 weeks.
- MSB0010841 120 mg: MSB0010841 was administered at a dose of 120 mg as SC injection every other week for a total duration of 6 weeks.
- MSB0010841 240 mg: MSB0010841 was administered at a dose of 240 mg as SC injection every other week for a total duration of 6 weeks.
- Placebo: Placebo matched to MSB0010841 was administered as SC injection every other week for a total duration of 6 weeks.
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
percentage of subjects
  Day 8 | 0 | 38 | 13 | 11 | 0
  Day 15 | 25 | 25 | 13 | 56 | 0
  Day 22 | 50 | 50 | 50 | 67 | 0
  Day 29 | 63 | 63 | 88 | 78 | 0
  Day 36 | 63 | 88 | 75 | 67 | 0
  Day 43 | 75 | 88 | 75 | 67 | 0
  Day 50 | 75 | 88 | 100 | 89 | 0
  Day 85 | 88 | 88 | 88 | 100 | 0

42. Secondary Outcome: Mean Percent Change From Baseline in the Body Surface Area (BSA) Affected by Psoriasis at Day 8, 15, 22, 29, 36, 43, 50 and 85
Description: The BSA is the physician's evaluation for the extent of disease. The entire body area is divided into 4 districts: head, upper limbs, trunk and lower limbs to which corresponds the 10%, 20%, 30% and 40% of the entire body surface respectively. The investigator assesses the percentage of the subjects' body surface area affected by psoriasis in each district. The final affected BSA value is the sum of the percentage of each district.
Time Frame: Baseline, Day 8, 15, 22, 29, 36, 43, 50 and 85
Population: Safety analysis set included all 41 subjects who received at least 1 dose of IMP (MSB0010841 or placebo). Here "n" signifies those subjects who were evaluable for this outcome measure at the specified time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
percent change
  Change at Day 8 (n=8,8,8,8,8) | 0.4 (1.14) | -30.0 (31.23) | -13.7 (15.13) | -12.5 (23.81) | 2.9 (23.32)
  Change at Day 15 (n=8,8,8,8,8) | 0.4 (1.14) | -33.1 (35.97) | -20.5 (10.98) | -51.1 (43.17) | -4.2 (12.21)
  Change at Day 22 (n=8,8,8,8,8) | -11.6 (24.90) | -40.2 (40.68) | -42.6 (27.15) | -68.5 (38.71) | -5.1 (12.69)
  Change at Day 29 (n=8,8,8,8,8) | -22.6 (26.35) | -44.1 (42.53) | -55.9 (36.56) | -82.9 (34.46) | -0.1 (26.13)
  Change at Day 36 (8,8,7,7,7) | -31.4 (22.96) | -52.7 (37.57) | -64.6 (37.65) | -83.5 (31.60) | -0.5 (27.92)
  Change at Day 43 (8,8,8,9,8) | -52.6 (32.91) | -65.2 (28.61) | -75.4 (37.35) | -82.2 (36.64) | -1.5 (27.05)
  Change at Day 50 (n=8,8,8,9,8) | -56.2 (34.71) | -69.4 (25.85) | -79.1 (32.30) | -82.2 (36.64) | -10.0 (17.87)
  Change at Day 85 (8,8,8,9,8) | -60.4 (33.51) | -61.3 (33.89) | -82.1 (31.05) | -95.5 (11.02) | -13.0 (20.13)

43. Secondary Outcome: Percentage of Subjects With Exacerbation of Psoriasis
Description: Psoriasis exacerbation was defined as either a worsening of 25% over the baseline value of the PASI score (PASI score at any visit >=125% of baseline PASI).
Time Frame: Baseline up to Day 85
Population: Safety analysis set included all 41 subjects who received at least 1 dose of IMP (MSB0010841 or placebo).
Measure: Number; unit: percentage of subjects
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 8
percentage of subjects | 0 | 0 | 0 | 0 | 12.5

ADVERSE EVENTS:
Time Frame: Baseline up to Day 85
Arm/Group | MSB0010841 30 mg | MSB0010841 60 mg | MSB0010841 120 mg | MSB0010841 240 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 5/8 | 5/8 | 6/9 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB0010841 30 mg (N=8) | MSB0010841 60 mg (N=8) | MSB0010841 120 mg (N=8) | MSB0010841 240 mg (N=9) | Placebo (N=8)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSB0010841 30 mg (N=8) | MSB0010841 60 mg (N=8) | MSB0010841 120 mg (N=8) | MSB0010841 240 mg (N=9) | Placebo (N=8)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 1
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
As AUCextra was more than 20% of AUC0-inf after first dose, AUCextra and all values derived from λz were regarded as implausible and "AUC0-inf", "MRT0-inf", "t1/2", "λz", "CL/f", and "Vz/f" were not calculated after first dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No